CLINICAL TRIAL: NCT06565234
Title: A Prospective Observational Study on the Integration of Virtual and Augmented Reality in Neurosurgical Planning, Education, and Patient Engagement
Brief Title: VR in Neurosurgery: Planning, Training & Communication
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Attill Saemann, Principal Investigator, University Hospital, Basel, Switzerland
Other Study IDs: 2023-02009; ko23Guzman3
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Brain Pathology
Keywords: Intracranial Pathology; Cerebrovascular or Skull Base Pathologies; Neurosurgery; Virtual Reality; Virtual Reality-demonstration; Virtual Reality-assisted Informed Consent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This prospective study analyzes the broad impact of virtual reality (VR) assistance on aneurysm surgeries through two primary focuses: first, it evaluates VR-assisted clip planning by examining its clinical outcomes in the operative management of aneurysms, and second, it investigates the role of VR-assisted patient-informed consent, including its effects on patient comprehension, the patient-doctor relationship, and anxiety.

DETAILED DESCRIPTION:
Over the last years, increasing innovations and accessibility to virtual reality (VR) and augmented reality (AR) technologies have contributed to the relevance of these tools in daily life and medical research activities. Surgical specialties play a key role in introducing these technologies into clinical practice, with additional applications and research fields.

In neurosurgery, VR-based surgical planning for aneurysm management has shown the potential to enhance patient safety, reduce surgery times, and improve clinical outcomes. Recently, a few studies have shown that patients can also benefit from using VR applied to IC, although the current patient-oriented use of VR remains scarce.

With the increasing demand for concepts like shared decision-making and patient-centered care, optimal IC is more relevant than ever. A pilot study (NCT) on VR-based IC at the investigators' institution demonstrated feasibility and indicated positive outcomes based on the investigators' questionnaire. Building on these findings, this prospective study aims to evaluate the broad impact of VR assistance on aneurysm surgeries by focusing on two main aspects: VR-assisted clip planning, including its effects on patient safety, operative times, and clinical outcomes, and VR-assisted patient-informed consent, examining subjective patient comprehension, the patient-doctor relationship, and anxiety. Additionally, the study will assess the cost-benefit ratio and feasibility of VR-based approaches in a routine clinical setting. Ultimately, VR may foster a better understanding of complex procedures, optimize the perioperative process for both patient and surgeon, reduce anxiety, and improve patient safety.

ELIGIBILITY:
Inclusion Criteria:

* The patient is able to give written consent (or written consent by legal representative)
* Preoperative imaging demonstrating intracranial pathology
* Cognitively able to provide answers for the questionnaires

Exclusion Criteria:

* No informed consent
* Adult patients without the power of judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for cerebrovascular or skull base pathologies at the University Hospital Basel or the University Children's Hospital Basel and/or their respective caretakers.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Time for clip application | Day 1 (Surgery)
  Intraoperative timestampf for opening, dissection, aneurysm preparation, clip application and possible clip replacement
Virtual Reality-Questionnaire | Day 0 (before surgery), >Day 2, Week 4, and Month 6 (after surgery)
  To assess each patient's experience during the consent process, we use the Virtual Reality Questionnaire (VRQ). The VRQ is a numeric scale ranging from 0 (least positive experience) to 10 (most positive experience). Higher scores indicate a better (more positive) outcome in terms of the patient's overall experience. This questionnaire has been specifically customized for the study's focus on virtual reality-based interventions.
Shared Decision Making Questionnaire (SDM-Q-9) | Day 0 (before surgery), >Day 2, Week 4, and Month 6 (after surgery)
  To assess the individual experience in consenting of the patient, the Shared Decision Making Questionnaire (SDM-Q-9) is used. The SDM-Q-9 is a 9-item questionnaire designed to measure the extent of shared decision-making between patients and healthcare providers. Each item is scored on a 6-point scale from 0 (completely disagree) to 5 (completely agree). Higher scores reflect a greater involvement of the patient in the decision-making process, indicating better shared decision-making practices.
Beck Anxiety Inventory (BAI) | Day 0 (before surgery), >Day 2, Week 4, and Month 6 (after surgery)
  To assess the individual experience in consenting of the patient, the Beck Anxiety Inventory (BAI) is used. The BAI is a 21-item self-report questionnaire used to assess the severity of an individual's anxiety. Each item is rated on a 4-point scale from 0 (not at all) to 3 (severely, it bothered me a lot). Higher scores indicate higher levels of anxiety, with scores categorized into minimal, mild, moderate, and severe anxiety levels.
Quality of Recovery-15 (QoR-15) | Day 0 (before surgery), >Day 2, Week 4, and Month 6 (after surgery)
  To assess the individual experience in consenting of the patient, the Quality of Recovery-15 (QoR-15) is used. The QoR-15 is a 15-item questionnaire used to evaluate a patient's recovery after surgery. It covers various aspects of recovery, including physical comfort, emotional state, physical independence, psychological support, and pain. Each item is rated on an 11-point scale from 0 (none of the time) to 10 (all of the time), with higher scores indicating better quality of recovery.

SECONDARY OUTCOMES:
Resources required for 3D visualization | Day 0 (before surgery)
  To determine the resources required to construct the 3D model, information regarding the required time, imaging modalities, and hardware is collected.
Length of hospitalization | Up to week 1
  As a standard clinical parameter the length of hospitalization is determined.
Modified Rankin Scale (mRS) | >Day 2, Week 4, and Month 6 (after surgery)
  As a standard clinical parameter the Modified Rankin Scale (mRS) is assessed. The mRS is a measure used to evaluate the degree of disability or dependence in daily activities of people who have suffered neurological pathologies. The scale ranges from 0 to 6, with 0 indicating no symptoms, 1 indicating no significant disability despite symptoms, and higher scores indicating increasing levels of disability up to 5, which represents severe disability requiring constant care, and 6 indicating death. Lower scores indicate less disability, while higher scores reflect greater disability.
Extended Glasgow Outcome Scale (eGOSE) | >Day 2, Week 4, and Month 6 (after surgery)
  As a standard clinical parameter the Extended Glasgow Outcome Scale (eGOSE) is assessed. The eGOSE is used to assess the functional outcome of patients after a brain pathology. The scale ranges from 1 to 8, with 1 indicating death and 8 indicating an upper good recovery with the patient resuming normal activities without disability. Lower scores indicate more severe disability or worse outcomes, while higher scores reflect better functional recovery and less disability.
Clip Specifics | d0 (before surgery), d1 (surgery)
  Comparison of preoperatively planned clip and intraoperative applied clip. Clip type, length, clipping method, expectation of remnant or need for provisional clipping.

CONTACTS AND LOCATIONS:
Overall Officials: Attill Saemann, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland